CLINICAL TRIAL: NCT03727035
Title: Quantification of CD163 Inflammatory Biomarker in Subgingival Plaque Samples of Generalized Chronic Periodontitis With or Without Type II Diabetes Mellitus
Brief Title: Quantification of CD163 Inflammatory Biomarker in Chronic Periodontitis and Diabetic Subjects
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meenakshi Ammal Dental College and Hospital (Other)
Responsible Party: Principal Investigator, Dr.Jaideep Mahendra, Professor and PhD guide, Meenakshi Ammal Dental College and Hospital
Other Study IDs: MADC/IRB-XV/2017/302
Record Dates: First submitted 2018-10-30; First posted 2018-11-01 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Periodontal Diseases
Keywords: CD163, Chronic periodontitis
MeSH Terms: conditions — Periodontal Diseases; Chronic Periodontitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: Group I :40 Generalized chronic periodontitis subjects without type II diabetes mellitus
- Group II: Group II: 40 Generalized chronic periodontitis subjects diagnosed with type II diabetes mellitus

SUMMARY:
The quantification of CD163 will be analysed in the subgingival plaque samples of generalized chronic periodontitis patients with and without diabetes mellitus. The demographic and the periodontal parameters were assessed and the correlated with the quantification of the CD163. The CD163 gene expression was analyzed with RT-PCR and the quantification of CD163 will be done using ELISA.

DETAILED DESCRIPTION:
The quantification of CD163 will be analysed in the subgingival plaque samples of generalized chronic periodontitis patients with and without diabetes mellitus. A total of 80 subjects with generalized chronic periodontitis were selected and divided into two groups. Group I comprised of 40 subjects who were diagnosed with generalized chronic periodontitis without any systemic conditions. Group II comprised of 40 generalized chronic periodontitis patients with type II diabetes mellitus. Demographic variables such as age, weight, height, BMI and income and the clinical parameters such as plaque index, bleeding on probing, probing pocket depth and clinical attachment level were recorded. Subgingival plaque samples were collected from both the groups.The collected samples were subjected to further molecular analysis for the CD163 expression using RT-PCR and for the CD163 quantification using ELISA. The elevated levels of CD163 in the subgingival plaque samples of generalized chronic periodontitis subjects with diabetes is expected and the early identification of patients at risk for diabetes mellitus and periodontitis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients willing to participate in the study.
2. Patients within the age group of 30-65 years (both male and female)
3. Patients should have ≥ 10 natural teeth.
4. Criteria for selection of generalized chronic periodontitis:

   * Patients having 30% or more sites with clinical attachment loss(CAL) ≥ 5mm.
5. Criteria for selection of type II diabetes mellitus:

   * Patients having HbA1C <7

Exclusion Criteria:

1. Patients with systemic conditions such as respiratory diseases, renal disease, liver disease, rheumatoid arthritis, allergy, advanced malignancies and HIV infection will be excluded from the present investigation.
2. Patients on drugs such as corticosteroids, antibiotics, aspirin, within 3months of investigation will be excluded.
3. Current smokers, individuals who quit smoking less than 6 months.
4. Patients who had undergone periodontal therapy within the previous 6 months.
5. Pregnant women (which may alter the oral flora).

Ages: 30 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients within the age group of 35-60 years. The subjects were from the South Indian population.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-02-10 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
Expression of CD163 gene | 12 months
  Expression of CD163 gene using RT-PCR

SECONDARY OUTCOMES:
Quantify the levels of CD163 | 12 months
  Quantify the levels of CD163 using ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Jaideep Mahendra, MDS,PhD, Study Director — Meenakshi Ammal Dental College
Locations (1):
- Jaideep Mahendra, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Detzen L, Chen SCY, Cheng B, Papapanou PN, Lalla E. Increased levels of soluble CD163 in periodontitis patients. J Clin Periodontol. 2017 Jun;44(6):585-590. doi: 10.1111/jcpe.12731. Epub 2017 May 16. PMID 28419494